CLINICAL TRIAL: NCT06966869
Title: Pharmacokinetic Study Evaluating the Absorption of Fentanyl From Transdermal Patches in Hemodynamically Unstable Versus Stable Patients Admitted to the Surgical Intensive Care Unit.
Brief Title: Evaluation of Fentanyl Transdermal Patch Absorption in Hemodynamically Unstable ICU Patients.
Status: Recruiting | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TLV-0344-24
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Pain Management; Critical Illness
Keywords: Transdermal fentanyl; Critical illness; Hemodynamic instability
MeSH Terms: conditions — Agnosia; Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemodynamically stable ICU patients receiving transdermal fentanyl without norepinephrine
  Interventions: Drug: Transdermal fentanyl patch
- Hemodynamically unstable ICU patients receiving transdermal fentanyl and intravenous norepinephrine
  Interventions: Drug: Transdermal fentanyl patch

INTERVENTIONS:
Drug: Transdermal fentanyl patch — The fentanyl patch will be applied as per standard ICU protocol for pain management. Blood levels will be monitored every 4 hours for 48 hours. Patients in this group require norepinephrine (>5 drops/hour of 4 mg/50 mL) to maintain MAP ≥ 65 mmHg.
  Groups: Hemodynamically unstable ICU patients receiving transdermal fentanyl and intravenous norepinephrine
Drug: Transdermal fentanyl patch — The fentanyl patch will be applied as per standard ICU protocol for pain management. Blood levels will be monitored every 4 hours for 48 hours. Patients in this group maintain MAP ≥ 65 mmHg without norepinephrine infusion.
  Groups: Hemodynamically stable ICU patients receiving transdermal fentanyl without norepinephrine

SUMMARY:
This study investigates how well fentanyl is absorbed through the skin when delivered via a transdermal patch in critically ill surgical ICU patients. It compares hemodynamically stable patients with unstable patients who require vasopressors to maintain adequate blood pressure. Fentanyl blood levels will be measured over time to assess whether absorption is impaired in unstable patients. The goal is to determine whether transdermal fentanyl is a viable option for pain management in resource-limited ICUs or in situations where intravenous fentanyl is unavailable.

DETAILED DESCRIPTION:
This is a single-center, pharmacokinetic study evaluating fentanyl absorption from transdermal patches in critically ill patients admitted to the surgical intensive care unit (ICU). A total of 40 patients will be recruited and divided into two groups. Both groups will receive a transdermal fentanyl patch for pain management. The grouping is based on hemodynamic status: 20 patients will be classified as hemodynamically unstable, defined by the need for intravenous norepinephrine infusion (≥5 drops/hour of a 4 mg/50 mL solution) to maintain a mean arterial pressure (MAP) of at least 65 mmHg. The other 20 patients will be considered hemodynamically stable, maintaining a MAP ≥ 65 mmHg without norepinephrine infusion. Patients who require very high doses of norepinephrine (over 20 drops/hour), with or without vasopressin, will be excluded.

The objective is to determine whether hemodynamic instability affects the systemic absorption of fentanyl from transdermal patches. Blood levels of fentanyl will be measured every 4 hours for the first 48 hours following patch application. The area under the concentration-time curve (AUC) will be calculated for each participant. The primary outcome is the difference in AUC between the stable and unstable groups.

Secondary variables include clinical and physiological factors that may influence fentanyl absorption, such as age, sex, body mass index (BMI, as a proxy for adiposity), body temperature, and liver function.

To ensure appropriate pain control in all participants, supplemental analgesia (non-fentanyl-based) will be administered during the first 24 hours after patch application and again at 48-72 hours, as needed. The ICU nursing team will routinely assess pain using validated tools such as the Behavioral Pain Scale (BPS), in accordance with standard unit practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-70 years.
* Male or female patients.
* Admitted to the surgical intensive care unit (ICU).
* Indications for pain management using fentanyl.

Exclusion Criteria:

* No clinical indication for fentanyl analgesia (e.g., pain well controlled with non-opioid medications).
* Known allergy or hypersensitivity to fentanyl.
* Contraindications to fentanyl (e.g., severe constipation, hepatic failure)
* Patients infected with multidrug-resistant organisms require high-level isolation (biosafety level 2 or higher).
* Hemodynamically very unstable patients requiring >20 drops/hour of norepinephrine (4 mg/50 mL), with or without vasopressin support.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients admitted to a surgical intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2028-04-22 (Estimated); Study Completion 2028-04-22 (Estimated)

PRIMARY OUTCOMES:
Difference in fentanyl absorption (AUC) between stable and unstable ICU patients | From patch application to 48 hours post-application
  Comparison of the area under the fentanyl concentration-time curve (AUC) between hemodynamically unstable and stable ICU patients receiving a transdermal fentanyl patch. Blood samples will be taken every 4 hours over a 48-hour period following patch application.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel, Israel